CLINICAL TRIAL: NCT02718677
Title: NON-INTERVENTIONAL STUDY TO ASSESS THE HEALTH-RELATED QUALITY OF LIFE IN SEVERE OR MODERATELY SEVERE HEMOPHILIA A SUBJECTS TREATED WITH REFACTO AF ROUTINE PROPHYLAXIS
Brief Title: Patient-reported Outcomes in Subjects Treated With ReFacto AF Routine Prophylaxis
Status: Withdrawn | Type: Observational
Why Stopped: Company decision to not conduct study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1831088
Record Dates: First submitted 2016-02-22; First posted 2016-03-24 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; recombinant factor VIII SQ

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1. Refacto AF (NIS): Non-Interventional Study
  Interventions: Drug: Refacto AF

INTERVENTIONS:
Drug: Refacto AF — Observational - Non-Interventional Study
  Other Names: moroctocog alfa

SUMMARY:
This NIS aims to assess the patient-reported outcomes (PROs) in enrolled subjects

DETAILED DESCRIPTION:
The design of the study is observational: both prospective and retrospective, national, multicenter, non- interventional. During this observational study, subjects diagnosed with severe or moderately severe (with severe phenotype) hemophilia A receiving routine prophylaxis treatment with ReFacto AF as per local standard clinical care, and in line with local labeling, are to be observed for 12 months.

The primary objective is to assess the health-related quality of life in subjects treated with ReFacto AF routine prophylaxis at baseline and after 6 and 12 months.

The secondary objectives are:

* To assess the subjective physical functioning of subjects treated with ReFacto AF routine prophylaxis at baseline and after 6 and 12 months;
* To assess the treatment satisfaction of caregivers of children and subjects above 18 years treated with ReFacto AF routine prophylaxis at baseline and after 6 and 12 months;
* To determine in routine clinical practice the mean annualized bleeding rate (ABR) in subjects treated with ReFacto AF routine prophylaxis;
* To describe the status of joint health measured by HJHS before and after starting routine prophylaxis for subjects above 18 years.

ELIGIBILITY:
Inclusion Criteria:

1. Severe (FVIII: C <1%) or moderately severe (FVIII: C ≥1 - ≤2% with severe phenotype [at least 4 spontaneous bleeds clinically documented during a 6 months period] and without inhibitors) male subjects with hemophilia A receiving routine prophylaxis treatment.
2. Age:

   * From 2 to 18 years;
   * Subjects above 18 years who began routine prophylaxis treatment in childhood (and were part of the national prophylaxis program when turned 18 years).
3. Previously treated patients (PTPs) with hemophilia A. Previously treated patient (PTP) is considered in this study as a subject who has at least 50 exposure days to any FVIII product. An exposure day (ED) is a 24-hour period during which a dose of FVIII concentrate has been administered, irrespective of size and frequency.
4. No history and no current FVIII inhibitor defined as a titer ≥0.6 BU/mL or any measured Bethesda inhibitor titer greater than the upper limit of normal for the laboratory performing the assay.
5. Subjects who are scheduled by their treating physician to initiate prophylaxis with ReFacto AF or to continue previously initiated prophylaxis with ReFacto AF, and subjects who are switching from prophylaxis with another FVIII product to ReFacto AF.
6. Evidence of a personally signed and dated informed consent and assent (for children 6-17 years of age) document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Main Exclusion Criteria:

1. Subject has known hypersensitivity to the active substance or any of the excipients.
2. Subject has known allergic reaction to hamster proteins.
3. Presence of any bleeding disorder in addition to hemophilia A.
4. Treatment with any investigational agent or device within the past 30 days.
5. Any other contraindications according to Summary of Product Characteristics (SPC).
6. Unsuitable to participate in study for any other reason as assessed by the investigator.
7. Subjects (or a legally acceptable representative) not able to understand study documents and study procedure.

Ages: 2 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Subjects receiving routine prophylaxis treatment with ReFacto AF as determined by the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The health-related quality of life in subjects treated with ReFacto AF routine prophylaxis | Baseline and after 6 and 12 months.
  HRQoL will be assessed by applying the self-reported hemophilia-specific quality of life Haemo-QoL questionnaire.
  The endpoint will include the domains and total scores of the questionnaire. The results of this study will be presented using descriptive statistics and there will be no hypothesis testing. The domain scores and total scores will be summarized by: N, mean (sd), median, min-max and the 95% confidence interval at baseline, end of study, and the change from baseline.
The health-related quality of life | Baseline and after 6 and 12 months.
  HRQoL will be be evaluated also by recording the number of days of absence from kindergarten, school or high-school. There are no a priori hypotheses specified and results will be presented as descriptive statistics.

SECONDARY OUTCOMES:
The subjective physical functioning of subjects treated with ReFacto AF routine prophylaxis | Baseline and after 6 and 12 months;
  Subjects will be asked to report their subjective physical functioning using the HEP-Test-Q.
  The endpoint will include the domains and total scores of the questionnaire. The results of this study will be presented using descriptive statistics and there will be no hypothesis testing. The domain scores and total scores will be summarized by: N, mean (sd), median, min-max and the 95% confidence interval at baseline, end of study, and the change from baseline.
The treatment satisfaction of caregivers of children and subjects above 18 years treated with ReFacto AF routine prophylaxis | Baseline and after 6 and 12 months;
  Caregivers will evaluate their satisfaction with the treatment of their child and the above 18 years subjects will evaluate their own satisfaction with the treatment using the Hemo-Satp questionnaire.
  The endpoint will include the domains and total scores of the questionnaire. The results of this study will be presented using descriptive statistics and there will be no hypothesis testing. The domain scores and total scores will be summarized by: N, mean (sd), median, min-max and the 95% confidence interval at baseline, end of study, and the change from baseline.
The mean annualized bleeding rate (ABR) in subjects treated with ReFacto AF routine prophylaxis; | After 12 months
  ABR will be calculated at the end of the study based on the number of bleeds recorded during the 12-months observation period. The ABR will be presented as N, mean (sd), median, min-max and the 95% confidence interval.
Joint health for subjects above 18 years | After 12 months
  Status of joint health will be described for subjects above 18 years using the HJHS (Hemophilia Joint Health Score) before and after starting routine prophylaxis. HJHS for one particular joint (elbow, knee or ankle) represents the sum between the joint totals and the global gait score.The minimum score is 0 and the maximum is 24.
  The joint totals is the sum between the scores for swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain and strength; the maximum score is 20.
  The global gait score evaluates walking, stairs, running and hopping in one leg; the maximum score is 4.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831088&StudyName=Non-interventional%20Study%20To%20Evaluate%20Efficacy%20And%20Safety%20Of%20Refacto%20Af%20In%20The%20Standard%20Prophylaxis%20Treatment%20Of%20Children%20With%20Severe%20Hemophilia%20A